CLINICAL TRIAL: NCT03830788
Title: Erectile Dysfunction in Good Prognosis Prostate Cancer: a Phase III Medico-economic Study Comparing Brachytherapy to Stereotactic Body Radiotherapy
Brief Title: Erectile Dysfunction in Good Prognosis Prostate Cancer : Comparison Between Brachytherapy and Stereotactic Body Radiotherapy
Acronym: TEMPOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Center Eugene Marquis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-2-10-003
Record Dates: First submitted 2019-01-31; First posted 2019-02-05 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
Keywords: SBRT; brachytherapy; localized low-risk and intermediate risk prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brachytherapy (Active Comparator): radiation by brachytherapy: brachytherapy by Iodine 125 delivering 144 Gy to the prostate
  Interventions: Radiation: Radiation by brachytherapy
- stereotactic body radiotherapy (SBRT) (Experimental): radiation by SBRT: SBRT delivers 7.25 Gy per fraction, in five fractions, corresponding to a total dose of 36.25 Gy to the prostate. Fiducials are implanted in the prostate. The prostate can be tracked/localized/treated thanks to the Cyberknife or a conventional linac equipped with an ExacTrac or a Calypso4D system.
  Interventions: Radiation: Radiation by SBRT

INTERVENTIONS:
Radiation: Radiation by brachytherapy — Brachytherapy by Iodine 125 delivering 144 Gy to the prostate
  Arms: Brachytherapy
Radiation: Radiation by SBRT — SBRT delivers 7.25 Gy per fraction, in five fractions, corresponding to a total dose of 36.25 Gy to the prostate. Fiducials are implanted in the prostate.
  Arms: stereotactic body radiotherapy (SBRT)

SUMMARY:
The TEMPOS-GEniToUrinary Group (GETUG) study is a multicenter, medico-economic study comparing brachytherapy to SBRT in low and intermediate risk prostate cancer, particularly focused on the issue of erectile dysfunction. A total of 240 potent patients are randomized in two arms. The experimental arm consists of SBRT delivering 7.25 Gy per fraction, in five fractions, corresponding to a total dose of 36.25 Gy to the prostate. The control arm consists of brachytherapy by Iodine 125 delivering 144 Gy to the prostate. The main objective of this health economics study is to perform a cost-utility analysis of SBRT compared to "standard" Iodine 125 brachytherapy in low-risk prostate cancer, 3 years after treatment. The endpoint is the Incremental Cost-Utility Ratio (ICUR) between SBRT and brachytherapy as primary criterion, expressed in cost per quality adjusted life year (QALY) gained. Cost-effectiveness analyses are performed as secondary objective with Incremental Cost-Effectiveness Ratios (ICERs) expressed as cost per erectile dysfunction avoided and cost per Life Year Gained. A long term evaluation is also performed, including a cost-utility, cost-effectiveness and budget impact analysis at 5 years, a comprehensive assessment of the erectile dysfunction up to 5 years after treatment, an evaluation of acute and late genito-urinary (GU) and Gastro-Intestinal (GI) toxicities, and of quality of life up to 5 years after treatment.

Eight patients/year/center are expected to be recruited in 2 years in about twenty participating centers.

In total, to our knowledge, this study will be the first health economic evaluation which compares SBRT versus Iodine 125 brachytherapy in low risk and intermediate risk prostate cancer. Both cost-utility and cost-effectiveness analyses will also provide useful and complementary information to decision makers in order (i) to recommend the best strategy to adopt; (ii) to estimate the budget impact on the French National Health Insurance of the generalization of the cost-effective strategy. Finally, this study will allow to assess and compare accurately the erectile dysfunction after both treatment modalities.

ELIGIBILITY:
Main inclusion criteria

* Biopsy proven prostate adenocarcinoma,
* Low risk prostate cancer according to d'Amico (T1-T2a and PSA <10 ng/ml, and Gleason score 6) or intermediate risk prostate cancer according d'Amico but excluding tumor with Gleason score 7 (4 + 3),
* Indication of a curative treatment by brachytherapy validated in multidisciplinary consultation meeting,

Main exclusion criteria

* Androgen deprivation therapy,
* Contraindication for prostate Iodine 125 brachytherapy (Prostate volume > 50 cc, impossibility if general anesthesia).
* Contraindication for Resonance Magnetic Imagery (RMI) (claustrophobia, pacemaker)
* Participation to another research which could have an impact on the study treatment and the outcomes

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2019-10-04 (Actual); Primary Completion 2030-04-04 (Estimated); Study Completion 2031-04-04 (Estimated)

PRIMARY OUTCOMES:
Cost-utility analysis of SBRT compared to "standard" Iodine 125 brachytherapy | 3 years after treatment.
  The cost-utility analysis is expressed in cost per quality adjusted life year (QALY) gained.

SECONDARY OUTCOMES:
Cost-utility analysis of SBRT compared to "standard" iodine-125 brachytherapy | 5 years after treatment
  The cost-utility analysis is expressed in cost per quality adjusted life year (QALY) gained.
Cost-utility analysis of avoided erectile dysfunction cost | 3 and 5 years after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Renaud De Crevoisier, PR, Principal Investigator — Centre Eugène Marquis
Locations (20):
- France (20):
  - Clinique Claude Bernard, Albi
  - ICO Paul Papin, Angers
  - Institut Bergonié, Bordeaux
  - Polyclinique Bordeaux-Aquitaine, Bordeaux
  - CLCC Georges-François Leclerc, Dijon
  - Centre Amethys - Charlebourg - La Défense, La Garenne-Colombes
  - Centre de Cobalthérapie Hartman, Levallois-Perret
  - CH Lyon Sud, Lyon
  - Institut régional du Cancer de Montpellier, Montpellier
  - Institut Curie, Paris
  - Hôpital Lyon Sud, Pierre-Bénite
  - Institut Jean Godinot, Reims
  - Centre Eugene Marquis, Rennes
  - Centre d'oncologie et de radiothérapie Saint Jean, Saint-Doulchard
  - Institut de Cancérologie de l'Ouest - Site Gauducheau, Saint-Herblain
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Institut Claudius Régaud, Toulouse
  - CHU Tours - Hôpital Bretonneau, Tours
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No